CLINICAL TRIAL: NCT01313156
Title: Lipids and Glucose Under Prospective Surveillance
Brief Title: LUPS-Lipids and Glucose Under Prospective Surveillance
Acronym: LUPS
Status: Completed | Type: Observational
Sponsor: Asklepios proresearch (Industry)
Collaborators: City of Hamburg (Other Government); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: AKS#1833
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2018-04

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes
Keywords: Metabolic Syndrome, Syndrome X, MetS,; Type 2 Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, non-randomized cohort study to analyse genetic variations, dietary patterns, perceived stress and anxiety and early changes in lipid metabolism leading to the metabolic syndrome and type 2 diabetes

DETAILED DESCRIPTION:
The LUPS-study is a collaboration between Asklepios Clinics Hamburg GmbH and University Clinic Hamburg Eppendorf, Germany. This study is assessing a multitude of serum biomarkers, anthropometrics, dietary habits, physical activity, perceived stress along with genetic information from "healthy workers" (25-60years) to better understand phenotype-genotype associations leading to MetS and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 25-60 years men and women willing to give consent

Exclusion Criteria:

* diabetes (type 1 or 2)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: so-called "Healthy-Workers", aged 25-60years, of Lufthansa-Technik, Hamburg, Germany, who voluntarily aggreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1962 (Actual)
Dates: Start 2008-11; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome, Type 2 Diabetes | 10 years
  assessing risk factors, e.g. HDL, BMI, Blood Pressure, FPG

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Mueller-Wieland, Prof., MD, Principal Investigator — Asklepios Klinik St.Georg, Hamburg, Germany; Karl Wegscheider, Prof., PHD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Germany
Locations (2):
- Germany (2):
  - Asklepios Klinik St.Georg, Hamburg
  - Universitätsklinikum Eppendorf, Hamburg

REFERENCES:
- [Derived] Muller-Wieland D, Altenburg C, Becher H, Burchard J, Frisch A, Gebhard J, Haas J, Harth V, Heeren J, Hengelbrock J, von Karais M, Knebel B, Kotzka J, Lowe B, Marx N, Pinnschmidt H, Preisser A, Rose M, Sawitzky-Rose B, Scheja L, Terschuren C, Toller M, Vettorazzi E, Wegscheider K. Development of the Metabolic Syndrome: Study Design and Baseline Data of the Lufthansa Prevention Study (LUPS), A Prospective Observational Cohort Survey. Exp Clin Endocrinol Diabetes. 2020 Dec;128(12):777-787. doi: 10.1055/a-0767-6361. Epub 2018 Nov 26. PMID 30477037